CLINICAL TRIAL: NCT07154888
Title: Fast Track to Fertility: Randomized Controlled Quality Improvement Initiative of an Algorithmic Text Messaging Communication and Patient Education Platform Designed to Improve the Efficiency the Fertility Workup
Brief Title: Fast Track to Fertility
Acronym: FTFRCT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FTFRCT
Record Dates: First submitted 2025-06-30; First posted 2025-09-04 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Infertility
Keywords: infertility; text messaging; patient education
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fast Track to Fertility Algorithmic Text Messaging Platform (Experimental): Patients randomized to the FTF arm will have a personalized algorithm selected on the W2H platform to send text messaging prompts about the next steps and provide educational materials. Patients in this arm will also receive text links to educational videos on the following subjects:
  * Diagnostic testing
  * Fertility awareness methods
  * Menstrual cycle
  * Optimizing natural fertility
  * Nutrition
  * Lifestyle modifications
  * Supplements
  * COVID and fertility
  * Mental health and fertility
  Interventions: Other: Fast Track to Fertility Algorithmic Text Messaging Platform
- Standard of Care (No Intervention): Patients randomized to the standard of care receive printed and/or electronic information about diagnostic tests and infertility treatments. A link to all video patient educational materials is included in this printed/electronic information. These educational materials will be provided at the first patient visit.

INTERVENTIONS:
Other: Fast Track to Fertility Algorithmic Text Messaging Platform — The Fast Track to Fertility algorithmic text messaging platform uses branching logic based on our standard workup protocol to text patients to schedule blood tests and an ultrasound timed to their menstrual cycle, as well as remind male partners to schedule blood and semen analyses.
  The platform will use an algorithmic approach to facilitate two-way communication, and any queries with no available responses will be escalated to the clinical team. Patients are not dependent on structured messages to progress through their journey; they can ask relevant questions in real time, and they are supported with fewer reminders. Response categories include clinical guidance and FAQs (e.g., how to determine cycle start or uterine cavity evaluation pre-appointment instructions), administrative guidance and FAQs (when to schedule test/appointment or clinic locations or phone numbers), and conversational pleasantries.
  Arms: Fast Track to Fertility Algorithmic Text Messaging Platform

SUMMARY:
The Fast Track to Fertility (FTF) program is an algorithmic text messaging communication and patient education platform designed to improve the efficiency the fertility workup. The initial pilot program resulted in an approximately 50% reduction in the time taken to complete the diagnostic workup. Since the pilot program, the investigators have enhanced the FTF Program (v2.0) beyond the texting platform, incorporating educational videos to increase patient knowledge and autonomy in the workup and treatment of infertility. This protocol pertains to a randomized controlled quality improvement initiative to measure the impact of the FTF v2.0 Program on fertility workup completion, efficiency, and patient outcomes.

DETAILED DESCRIPTION:
Infertility, recognized as a disease by the WHO, is defined as the failure to achieve successful pregnancy after at least 12 months of regular unprotected intercourse in women younger than age 35, or within 6 months in women 35 or older. The worldwide prevalence of infertility is high, affecting approximately 12-18% of couples. Through detailed medical history for risk factors, assessment of ovulatory function, structure and patency of the female reproductive tract, and semen analysis of the male partner, the cause of infertility can be ascertained in most patients and allows determination of appropriate therapeutic options.

Despite the high prevalence of infertility, only a small proportion of patients seek care, and an even smaller number continue care after the initial evaluation. Several studies have examined underlying reasons for early discontinuation of infertility care, namely prior to initiation of treatment. In a study from the Netherlands examining drop-out rates at different stages of fertility care, nearly half of the patients who discontinued care withdrew before initiating any treatment; 6.0% did not return after the first visit, 3.4% dropped out during the diagnostic work-up, and 35.7% dropped out after finishing the diagnostic workup. In a cohort of 434 infertile couples residing in urban United States, Eisenberg et al found that 13% did not pursue any infertility treatment after the initial consultation with a reproductive endocrinologist. When compared to patients pursuing treatment, these patients were typically older, less educated, of lower socioeconomic status, and had a higher baseline depression score. Of note, psychological factors are associated with higher drop-out rates even in patients with insurance coverage for infertility treatments. This data highlights that the initial evaluation and diagnostic work-up process is a critical stage of fertility care that engages patients and influences their decision to pursue treatment.

Although the barriers to pursuing fertility treatments have been studied, there is less information on the precise barriers to completing the diagnostic work-up. This first step can be cumbersome as it includes laboratory tests and radiographic or ultrasound imaging to evaluate the fallopian tube patency and uterine cavity in the female partner, blood tests and semen analysis in the male partner, and more recently, genetic carrier screening in both partners. What adds to the complexity of this testing is the need for time-sensitive and menstrual-cycle dependent testing which is required for the physician to recommend a personalized treatment plan. Poor communication or lack of understanding of the instructions can lead to missed testing windows, especially follicular phase appointments for blood tests and imaging studies. From a patient's perspective, each month that passes represents a missed opportunity to become pregnant further contributing to the higher levels of anxiety and stress associated with infertility diagnosis.

Based on contextual inquiry and grounded in patient needs, the work-up period was identified as an opportunity to optimize patient interactions with their physician. It was hypothesized that the implementation of a novel digital health platform to improve communication with patients regarding their diagnostic work-up will improve completion rates and overall patient retention. To this effect, the Fast Track to Fertility (FTF) program was created, which was developed using AI and natural language processing (NLP) to accurately provide semi-automated two-way text message communications to send reminders regarding the timing of tests, location of testing sites, and related educational materials. A detailed description of the discovery, pilot, and semi-automation phases of this innovative program has been published previously. A text-based approach was selected as it does not require downloading an app, supports real-time two-way engagement in a private setting, and has been shown to reduce racial disparities in care for reproductive-age women in our department.

The initial pilot program coupled with the iterative development phases resulted in an approximately 50% reduction in the time taken to complete the fertility work-up (from 97 days to 41 days) with high patient net promoter scores (>70%). In addition, high patient willingness to participate in this program (70%) and high accuracy of the AI-augmented texting (up to 80%) was observed, resulting in workflow improvement for staff and providers. However, it is not clear if these favorable outcomes were at least in part related to selection bias, as patients had to opt into the program and were not randomized. A secondary analysis on the barriers to infertility workup completion demonstrated that more Black women and those without fertility benefits both declined to enroll in the FTF program and did not initiate the infertility workup.

The goal of this proposed quality improvement initiative is to perform a randomized controlled quality improvement study on the updated FTF program (FTF v2.0). Since the initial pilot study was published, the FTF Program has been reworked. The platform now uses an algorithmic approach to text messaging (rather than AI) and incorporates several educational videos to increase patient knowledge and autonomy in the workup and treatment of infertility. Through this initiative, the aim is to measure the impact of the FTF program on infertility workup completion, fertility treatment initiation, pregnancy, and live birth.

ELIGIBILITY:
Inclusion Criteria:

* Female new patients seen at Penn Fertility Care for the workup of infertility
* Patients who have yet to complete at least 3 components of the fertility workup, including:

  1. Laboratory blood tests
  2. Tubal patency testing / uterine cavity assessment (hysterosalpingogram (HSG) or sonohysterogram (Femvue))
  3. Pelvic ultrasound
  4. Semen analysis
  5. Genetic carrier screening.
* Patients must be willing to be randomized to FTF versus standard of care

Exclusion Criteria:

* Pregnancy
* Age <18 years
* Patients with no access to texting or unable to engage via a text messaging service
* Patients requiring fewer than three components of the infertility work-up
* Patients presenting for second opinion with work-up completed
* Patients seeking IVF for oocyte cryopreservation, PGT-M, or embryo banking
* Non-English speaking

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-04-25 (Actual); Primary Completion 2025-10-22 (Actual); Study Completion 2027-04-25 (Estimated)

PRIMARY OUTCOMES:
Infertility workup completion | 60 days
  Number of subjects that completed all components of their personalized work-up with 60 days of the new patient visit

SECONDARY OUTCOMES:
Days taken to complete the infertility workup | One year following participant recruitment
Days between new patient and return visit | One year following participant recruitment
Percentage of patients who completed 3, 4, or 5 components of the work-up | One year following participant recruitment

OTHER OUTCOMES:
Number of patients initiating any fertility treatment | One year following participant recruitment
Number of patients specifically initiating IVF | One year following participant recruitment
Time to initiate fertility treatment | One year following participant recruitment
Time to initiate IVF | One year following participant recruitment
Number of pregnancies and live births over a one-year follow up period. | One year following participant recruitment

CONTACTS AND LOCATIONS:
Overall Officials: Anuja Dokras, MD, MHCI, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Penn Fertility Care, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The IPD that will be shared includes de-identified individual-level data related to primary and secondary outcome measures and baseline characteristics.
Supporting Information: Study Protocol, SAP
Time Frame: The data will be made available beginning 6 months after publication and will be accessible for 2 years.
Access Criteria: Data will be shared with qualified researchers upon request and with appropriate data use agreements. Interested researchers must submit a proposal outlining the research question and analysis plan.

REFERENCES:
- [Background] Acker A, Senapati S, Dokras A. Barriers to access: findings from an implementation study of an artificial intelligence-augmented 2-way chatbot for fertility care. Fertil Steril. 2023 Jul;120(1):199-201. doi: 10.1016/j.fertnstert.2023.04.016. Epub 2023 Apr 20. No abstract available. PMID 37085095
- [Background] Hirshberg A, Sammel MD, Srinivas SK. Text message remote monitoring reduced racial disparities in postpartum blood pressure ascertainment. Am J Obstet Gynecol. 2019 Sep;221(3):283-285. doi: 10.1016/j.ajog.2019.05.011. Epub 2019 May 20. No abstract available. PMID 31121137
- [Background] Lerma K, Reyes G, Tiwari S, Tewari A, Hastings C, Blumenthal PD. Acceptability of a text message-based fertility awareness application for family planning in Lucknow, India. Int J Gynaecol Obstet. 2018 Jul;142(1):104-107. doi: 10.1002/ijgo.12488. Epub 2018 Apr 6. PMID 29574716
- [Background] Senapati S, Asch DA, Merchant RM, Rosin R, Seltzer E, Mancheno C, et al. The Fast Track to Fertility Program: Rapid Cycle Innovation to Redesign Fertility Care. NEJM Catalyst 2022;3(10):CAT.22.0065.
- [Background] Fallahzadeh H, Zareei Mahmood Abadi H, Momayyezi M, Malaki Moghadam H, Keyghobadi N. The comparison of depression and anxiety between fertile and infertile couples: A meta-analysis study. Int J Reprod Biomed. 2019 May 5;17(3):153-62. doi: 10.18502/ijrm.v17i3.4514. eCollection 2019 Mar. PMID 31435599
- [Background] Domar AD. Impact of psychological factors on dropout rates in insured infertility patients. Fertil Steril. 2004 Feb;81(2):271-3. doi: 10.1016/j.fertnstert.2003.08.013. PMID 14967355
- [Background] Eisenberg ML, Smith JF, Millstein SG, Nachtigall RD, Adler NE, Pasch LA, Katz PP; Infertility Outcomes Program Project Group. Predictors of not pursuing infertility treatment after an infertility diagnosis: examination of a prospective U.S. cohort. Fertil Steril. 2010 Nov;94(6):2369-71. doi: 10.1016/j.fertnstert.2010.03.068. Epub 2010 May 14. PMID 20471010
- [Background] Brandes M, van der Steen JO, Bokdam SB, Hamilton CJ, de Bruin JP, Nelen WL, Kremer JA. When and why do subfertile couples discontinue their fertility care? A longitudinal cohort study in a secondary care subfertility population. Hum Reprod. 2009 Dec;24(12):3127-35. doi: 10.1093/humrep/dep340. Epub 2009 Sep 26. PMID 19783833
- [Background] Thoma ME, McLain AC, Louis JF, King RB, Trumble AC, Sundaram R, Buck Louis GM. Prevalence of infertility in the United States as estimated by the current duration approach and a traditional constructed approach. Fertil Steril. 2013 Apr;99(5):1324-1331.e1. doi: 10.1016/j.fertnstert.2012.11.037. Epub 2013 Jan 3. PMID 23290741
- [Background] Practice Committee of the American Society for Reproductive Medicine. Electronic address: asrm@asrm.org; Practice Committee of the American Society for Reproductive Medicine. Fertility evaluation of infertile women: a committee opinion. Fertil Steril. 2021 Nov;116(5):1255-1265. doi: 10.1016/j.fertnstert.2021.08.038. Epub 2021 Oct 2. PMID 34607703
- [Background] Practice Committee of the American Society for Reproductive Medicine. Electronic address: asrm@asrm.org. Definitions of infertility and recurrent pregnancy loss: a committee opinion. Fertil Steril. 2020 Mar;113(3):533-535. doi: 10.1016/j.fertnstert.2019.11.025. Epub 2020 Feb 27. PMID 32115183
- [Background] Zegers-Hochschild F, Adamson GD, de Mouzon J, Ishihara O, Mansour R, Nygren K, Sullivan E, Vanderpoel S; International Committee for Monitoring Assisted Reproductive Technology; World Health Organization. International Committee for Monitoring Assisted Reproductive Technology (ICMART) and the World Health Organization (WHO) revised glossary of ART terminology, 2009. Fertil Steril. 2009 Nov;92(5):1520-4. doi: 10.1016/j.fertnstert.2009.09.009. Epub 2009 Oct 14. PMID 19828144